CLINICAL TRIAL: NCT00169715
Title: Percutaneous Surgical Outcomes and Metabolic Findings in Patients With Stone-Bearing Calicial Diverticula
Brief Title: Database and Registry for Renal Diverticulum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana Kidney Stone Institute (Other)
Collaborators: University of Chicago (Other)
Responsible Party: James Lingeman, M.D., Methodist Urology, Indiana Kidney Stone Instititue
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 03-019
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Kidney Stones; Renal Calculi; Tic
Keywords: Kidney stones; renal Calculi; Tic; Caliceal Diverticula
MeSH Terms: conditions — Kidney Calculi; Tics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other)
  Interventions: Procedure: Percutaneous Caliceal Diverticuli

INTERVENTIONS:
Procedure: Percutaneous Caliceal Diverticuli — Standard of care to remove a stone from a caliceal diverticulum is to do a percutaneous procedure for stone removal and then fulgerate the diverticulum to prevent stone recurrence. We plan to aspirate urine from this diverticulum and compare it to urine collected from the renal pelvis of the same kidney.

SUMMARY:
Historically, percutaneous treatment of stone-bearing caliceal diverticula has resulted in the best success rates when examining factors such as symptom relief and stone-free rates (Jones, et al, 1991). Many groups have reported modifications in their percutaneous approach which have reportedly improved patient outcomes, but these series have very limited populations. Another issue concerning stone-bearing caliceal diverticula centers on the etiology of stones formation within these areas. This topic remains a subject of debate, with conflicting data in the literature.

DETAILED DESCRIPTION:
Caliceal diverticula are non-secretory cavities which are connected to the remainder of the renal collecting system through narrow infundibulae. Calculi are associated with these cavities from 9.5 to 78% of cases (Liatsikos, et al 2000; Monga, et al 2000). This subset of stone-forming patients often presents with recurrent urinary tract infections and flank discomfort. The definitive treatment for this entity remains surgical, with shock wave lithotripsy (SWL), ureteroscopy (URS), percutaneous nephrolithotomy (PNL), and laparoscopy all serving as management options. However, multiple groups have demonstrated that PNL remains the treatment modality of choice secondary to its superior stone-free and symptom relief rates (Jones, et al 1991; Donnellan, et al 1999; Shalhav, et al 1998). Over time, technique modifications have been reported by other groups (Monga, et al 2000; Auge, et al 2002) involving different methods of managing the infundibulum that connects the diverticulum to the rest of the renal collecting system. Our own surgical experience with percutaneous treatment of stone-bearing caliceal diverticula has resulted in various technique modifications as well, which we believe have continued to improve patient outcomes. To support our hypothesis, we will need to perform a systematic review our patient population to document these surgical outcomes.

Another question surrounding this subset of patients involves the primary factor responsible for the formation of calculi within the diverticula. Unfortunately, the literature has provided conflicting data on this issue. Some groups attribute stone formation to underlying metabolic abnormalities (Hsu, et al 1998). Other groups have not found any metabolic problems, instead concluding that impaired urinary drainage from the diverticulum primarily contributes calculus formation (Liatsikos, et al 2000). By prospectively obtaining urines on our caliceal diverticula patients, we hope that detailed metabolic analyses will allow us to conclude definitively whether metabolic abnormalities are prevalent in this population.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female patients over the age of 18 with symptomatic caliceal diverticular stone(s) who have had or require percutaneous treatment

EXCLUSION CRITERIA:

1. Patients unable to give informed consent
2. Patients with active bleeding diatheses
3. Women who are pregnant or in whom pregnancy status cannot be confirmed
4. Patients with renal insufficiency requiring dialysis
5. Patients with a baseline serum creatinine of 1.4 or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2003-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
We hope to use the urine metabolic data to clarify whether this subset of stone forming patients have significant underlying metabolic risk factors that contribute to stone formation within their diverticula. | Two months post-op

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — Methodist Urology, LLC
Locations (1):
- Methodist Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Kim SC, Kuo RL, Tinmouth WW, Watkins S, Lingeman JE. Percutaneous nephrolithotomy for caliceal diverticular calculi: a novel single stage approach. J Urol. 2005 Apr;173(4):1194-8. doi: 10.1097/01.ju.0000152320.41995.c2. PMID 15758742